CLINICAL TRIAL: NCT02000284
Title: Defining Subgroups of Mitochondrial Disease and Dysfunction in Autism Spectrum Disorder
Brief Title: Mitochondrial Dysfunction in Autism Spectrum Disorder
Acronym: Mito
Status: Active, not recruiting | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: Jane Botsford Johnson Foundation (Unknown); Arkansas Biosciences Institute (Unknown); The University of Texas Health Science Center at San Antonio (Other); St. Christopher's Hospital for Children (Other); The BRAIN Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 137162
Record Dates: First submitted 2013-11-21; First posted 2013-12-04 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder; Autism; Mitochondrial Disease; Developmental Delay
Keywords: Autism Spectrum Disorder; ASD; Autism; Pervasive developmental disorder - Not Otherwise Specified; PDD-NOS; Asperger's Syndrome; Mitochondrial Disease; Developmental Delay; Typical Development
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Mitochondrial Diseases; Learning Disabilities; Asperger Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biochemical Measures
  1. Mitochondrial Energetics
  2. Redox Metabolism
  3. ATP Measurement
  4. Mitochondrial Copy Number
  5. Clinical Laboratory Testing
  6. Urine Testing
  7. Stool Testing
  8. Teeth Collection
  9. Saliva Collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- General ASD: 150 general ASD children
- ASD/MD: 50 children Diagnosed with an Autism Spectrum Disorder and a Mitochondrial Disorder
- ASD/noMD: 50 children with ASD that have been r/o as having a mitochondrial disorder
- MD/noASD: 50 children with a mitochondrial disorder and without an ASD
- Developmental Delay: 50 children without a mitochondrial disorder or autism spectrum disorder, but with general developmental delays
- Typically Developing: 100 children with no history of medical, behavioral, or immunological disorders

SUMMARY:
Researchers at Arkansas Children's Hospital Research Institute are conducting a study about mitochondrial function in children. The study involves up to 5 visits to Arkansas Children's Hospital with fasting blood draws, behavioral assessments, and/or questionnaires.

This study is not currently recruiting, but continues to follow those who were enrolled.

There is no cost for visits or study-related exams.

For further information, please contact the program manager, Leanna Delhey, at ldelhey@uams.edu or 501-364-4519

DETAILED DESCRIPTION:
Objective: The main objective of this proposal is to develop a minimally-invasive biological assay that can be widely used to identify variations in mitochondrial function and dysfunction in children with autism spectrum disorder (ASD). This assay will allow the investigators to determine the true range of mitochondrial function and dysfunction across a population of children with ASD. The relationship between mitochondrial function and dysfunction in ASD, redox metabolism and core ASD symptomology will also be investigated. To understand the true variation in mitochondrial function and its relationship to cognitive development and autism symptoms, participants will be evaluated at two time points to understand the within subject variation of mitochondrial measurements.

Specific Aims: 1) To develop a minimally-invasive assay that can accurately identify children with ASD/MD from the general ASD population. 2) To establish whether there is simply an ASD/MD subgroup or whether mitochondrial dysfunction occurs on a spectrum from mild to severe in ASD. 3) To determine the relationship between mitochondrial function and redox metabolism in children with ASD. 4) To evaluate the effect of mitochondrial dysfunction and glutathione redox status on language and social development and ASD symptoms.

Study Design: Using the Seahorse Analyzer, investigators will develop profiles of mitochondrial function for individuals with ASD and known MD (ASD/MD) and individuals with ASD known not to have MD (ASD/NoMD). These two groups will serve as the two ends of the spectrum of mitochondrial function in children with ASD and will be compared to profiles from TD children. Investigators will then examine the profiles of mitochondrial function in a general population of individuals with ASD to determine how these individuals fall into this spectrum defined by the ASD/MD and ASD/NoMD groups, as well as DD and no ASD/MD. Glutathione redox metabolism will be measured in all participants. The relationship between mitochondrial function, redox metabolism and core ASD symptoms will be studied in the ASD groups with particular attention to whether ASD symptoms, language ability and adaptive behavior are directly related to mitochondrial function or indirectly related to mitochondrial function through its effect on redox metabolism.

Study Population: Investigators will recruit several groups of children for this study: 50 children with ASD who have MD (ASD/MD); 50 children with ASD who do not have MD (ASD/NoMD); 50 no ASD/MD; 50 no ASD/no MD but DD; 100 TD controls; and a general population of 150 children with ASD.

Children with ASD with and without MD will be identified in the autism multispecialty clinic (AMC), as well as the ATN and other medical clinics that evaluate children with ASD in outpatient clinics in Arkansas. When a child is identified, the study coordinator will contact the parents and describe the study. If the parents are interested, the coordinator will screen by asking inclusion/exclusion criteria questions. If the child qualifies, the coordinator will schedule the visit and mail consent forms to the parents for their review. During the visit they will undergo a blood draw for metabolic testing. The child will then be sent to breakfast since the blood tests require collection prior to breakfast. After breakfast the participant will undergo further language and behavioral assessment while the parent will be interviewed for the Vineland and other questionnaires. The parents will be provided questionnaires for the teacher to fill out and mail in an addressed, postage paid envelope.

For the TD participants, these children will be recruited in several ways including using social media through Arkansas Children's Hospital, flyers posted in the community (i.e. primary pediatric clinics), as well as referrals from pediatricians. When a child is identified, the study coordinator will contact the parents and describe the study. If the parents are interested, the coordinator will screen by asking inclusion/exclusion criteria questions. If the child qualifies, the coordinator will schedule the visit and mail consent forms to the parents for their review. During the visit they will undergo a blood draw for metabolic testing.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for ASD children

1. Autism Spectrum Disorder (As defined by a gold standard measure for ASD diagnosis: the Autism Diagnostic Observation Schedule, Autism Diagnostic Interview, and/or the minimum Arkansas state requirement for autism classification, as defined by a consensus diagnosis of ASD by a medical doctor, speech pathologist, and psychologist.). In an event where sufficient diagnostic information is lacking, and the PI believes that the clients meet all other inclusion criteria and a prospective diagnosis of an ASD is clinically warranted, and a formal diagnosis is scheduled to occur within a reasonable time frame from the date of study entry, then the client may be considered as potentially eligible.
2. 0 years through 17 years 11 months of age

Inclusion Criteria for TD children

1. 0 years to 17 years 11 months of age

Exclusion Criteria:

* Discussed on a case by case basis

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will recruit several groups of children for this study: 50 children with ASD who have MD (ASD/MD); 50 children with ASD who do not have MD (ASD/NoMD); 50 no ASD/MD; 50 no ASD/no MD but DD; 100 TD controls; and a general population of 150 children with ASD.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2012-10-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial Reserve Capacity measured using the Seahorse XR Flux Analyzer | up to one year
  Children with ASD will be differentiated from all other cohorts and have a specific pattern of mitochondrial dysfunction that will be different from and comparable to other groups of children in the study (e.g. mitochondrial disease without autism, typically developing, autism with mitochondrial disease, and developmental delay). It is hypothesized that these children will have a more pronounced delay in their development and will have a higher probability for poor developmental and behavioral outcomes. This will be evaluated using a Seahorse VR flux analyzer to generate a maximal reserve capacity value.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Rose, PhD, Principal Investigator — The University of Tennessee Health Science Center
Locations (1):
- The University of Tennessee Health Science Center, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Frye RE, Lionnard L, Singh I, Karim MA, Chajra H, Frechet M, Kissa K, Racine V, Ammanamanchi A, McCarty PJ, Delhey L, Tippett M, Rose S, Aouacheria A. Mitochondrial morphology is associated with respiratory chain uncoupling in autism spectrum disorder. Transl Psychiatry. 2021 Oct 13;11(1):527. doi: 10.1038/s41398-021-01647-6. PMID 34645790
- See also: Related Info — http://achri.archildrens.org/Clinical_Research/Studies/MitochondrialDiseaseASD.html

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT02000284/Prot_SAP_000.pdf